CLINICAL TRIAL: NCT06350513
Title: The Effect of Animated Film and Storybook on Fear and Anxiety Levels in Children With Newly Diagnosed Type 1 Diabetes: Randomized Controlled Study
Brief Title: The Effect of Animated Movies and Storybooks on Fear and Anxiety Levels in Children With Type 1 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selverhan Yurttutan (Other)
Responsible Party: Sponsor-Investigator, Selverhan Yurttutan, reserch asistant, Necmettin Erbakan University
Organization: Necmettin Erbakan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NecmettinE
Record Dates: First submitted 2024-03-15; First posted 2024-04-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Diabetes Mellitus, Type 1; Child, Only; Anxiety; Fear; Nurse
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Parallel Group (Experiment-Control) Randomized Controlled Experimental
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Animation movie, story book (Experimental): Animation movie: For this study, an animated film (Professor bumblebee animation) prepared for newly diagnosed children with type 1 diabetes will be shown in the experimental group. This is an approximately 10 minute film produced by Life for a children's center in New South Wales (DIABETES AUSTRALIA). The animated film will be translated into Turkish and sent to experts (specialists in the field of Children and Diabetes) for expert opinion. It will be shown to children after all permissions have been obtained following expert opinions. This animated movie is a guide to diabetes for children. Additionally, the storybook will be given as a gift for the children in the experimental group to read.
  Story Book: It is an educational booklet version of the Professor Bumblebee animation translated into Turkish and illustrated. The aim here is to serve as an auxiliary tool for newly diagnosed T1D children to look at later and where they are confused.
  Interventions: Other: Animation movie, story book
- control group (Other): No applications will be made.
  Interventions: Other: Animation movie, story book

INTERVENTIONS:
Other: Animation movie, story book — Animation movie: For this study, an animated film (Professor bumblebee animation) prepared for newly diagnosed children with type 1 diabetes will be shown in the experimental group. This is an approximately 10 minute film produced by Life for a children's center in New South Wales (DIABETES AUSTRALIA). The animated film will be translated into Turkish and sent to experts (specialists in the field of Children and Diabetes) for expert opinion. It will be shown to children after all permissions have been obtained following expert opinions. This animated movie is a guide to diabetes for children. Additionally, the storybook will be given as a gift for the children in the experimental group to read.
  Story Book: It is an educational booklet version of the Professor Bumblebee animation translated into Turkish and illustrated. The aim here is to serve as an auxiliary tool for newly diagnosed T1D children to look at later and where they are confused.

SUMMARY:
This study aims to evaluate the effects of animated films and story books on the fear and anxiety levels of children with newly diagnosed type 1 diabetes.

DETAILED DESCRIPTION:
This study aims to evaluate the effects of animated films and story books on the fear and anxiety levels of children with newly diagnosed type 1 diabetes. In the study, newly diagnosed children in the experimental group will be shown a 10-minute movie and read the educational booklet. Routine care will continue for the control group.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* Parental approval
* Being between the ages of 7-12,
* Being diagnosed with T1D for the first time,
* Being literate and able to communicate in Turkish

Exclusion Criteria:

* Having a mental, visual, hearing or communication impairment,
* Having mental and spiritual health problems,

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2024-02-25 (Actual); Primary Completion 2026-06-25 (Estimated); Study Completion 2026-07-25 (Estimated)

PRIMARY OUTCOMES:
State Anxiety Inventory for Children (STAI-C) | Initial assessment will be performed at baseline (pre-intervention)
  This scale was developed to evaluate children's state and trait anxiety and is in a self-report form. As a result of some procedures, the scale was turned into 2 separate scales containing a total of 40 items (20 state and 20 trait anxiety items). Although the validity and reliability of the scale has been done for children aged 9-12, the scale can be used until the age of 17 because it is difficult for children over the age of 12 to understand the adult anxiety scale. In the State Anxiety Scale for Children, children are asked to mark one of three options regarding how they evaluate how they feel at that moment. The scale aims to evaluate emotions related to state anxiety such as tension, irritability, rush, and uneasiness. The highest score that can be obtained from the State Anxiety Scale is 60 and the lowest score is 20. Cronbach's α value was found to be 0.82
State Anxiety Inventory for Children (STAI-C) | The second evaluation will be made after the first evaluation (after watching the animated movie and reading the story book (approximately 1 hour later)).
  This scale was developed to evaluate children's state and trait anxiety and is in a self-report form. As a result of some procedures, the scale was turned into 2 separate scales containing a total of 40 items (20 state and 20 trait anxiety items). Although the validity and reliability of the scale has been done for children aged 9-12, the scale can be used until the age of 17 because it is difficult for children over the age of 12 to understand the adult anxiety scale. In the State Anxiety Scale for Children, children are asked to mark one of three options regarding how they evaluate how they feel at that moment. The scale aims to evaluate emotions related to state anxiety such as tension, irritability, rush, and uneasiness. The highest score that can be obtained from the State Anxiety Scale is 60 and the lowest score is 20. Cronbach's α value was found to be 0.82
State Anxiety Inventory for Children (STAI-C) | The third evaluation will be made approximately 3 days after the second evaluation.
  This scale was developed to evaluate children's state and trait anxiety and is in a self-report form. As a result of some procedures, the scale was turned into 2 separate scales containing a total of 40 items (20 state and 20 trait anxiety items). Although the validity and reliability of the scale has been done for children aged 9-12, the scale can be used until the age of 17 because it is difficult for children over the age of 12 to understand the adult anxiety scale. In the State Anxiety Scale for Children, children are asked to mark one of three options regarding how they evaluate how they feel at that moment. The scale aims to evaluate emotions related to state anxiety such as tension, irritability, rush, and uneasiness. The highest score that can be obtained from the State Anxiety Scale is 60 and the lowest score is 20. Cronbach's α value was found to be 0.82

SECONDARY OUTCOMES:
Children's Fear Scale | Initial assessment will be performed at baseline (pre-intervention)
  The child fear scale was designed to measure a child's anxiety level and is intended to be used in children between the ages of 5-10. However, some suggest that it can also be used in children up to the age of 12. The child is shown five facial expressions (ranging from zero to four), each representing a level on the scale. Zero and four; Zero indicates no fear or anxiety, and four indicates high levels of fear and anxiety. This scale can be used to measure fear and anxiety before and during the procedure. Cohen's Kappa coefficient was checked to determine interobserver agreement.
Children's Fear Scale | The second evaluation will be made after the first evaluation (after watching the animated movie and reading the story book (approximately 1 hour later)).
  The child fear scale was designed to measure a child's anxiety level and is intended to be used in children between the ages of 5-10. However, some suggest that it can also be used in children up to the age of 12. The child is shown five facial expressions (ranging from zero to four), each representing a level on the scale. Zero and four; Zero indicates no fear or anxiety, and four indicates high levels of fear and anxiety. This scale can be used to measure fear and anxiety before and during the procedure. Cohen's Kappa coefficient was checked to determine interobserver agreement.
Children's Fear Scale | The third evaluation will be made approximately 3 days after the second evaluation.
  The child fear scale was developed by McMurtry et al. in 2011. The Turkish validity of the scale was determined by Gerçeker et al. It was made by in 2018. The child fear scale was designed to measure a child's anxiety level and is intended to be used in children between the ages of 5-10. However, some suggest that it can also be used in children up to the age of 12. The child is shown five facial expressions (ranging from zero to four), each representing a level on the scale. Zero and four; Zero indicates no fear or anxiety, and four indicates high levels of fear and anxiety. This scale can be used to measure fear and anxiety before and during the procedure. Cohen's Kappa coefficient was checked to determine interobserver agreement.

CONTACTS AND LOCATIONS:
Locations (3):
- Turkey (Türkiye) (3):
  - NecmettinEU, Konya, Meram
  - Semra Köse, Konya, Meram
  - Necmettin Erbakan Üniversity, Konya

IPD SHARING:
Plan to Share IPD: Yes